CLINICAL TRIAL: NCT02774083
Title: An Evaluation of the Feuerstein Instrumental Enrichment Program for the Cognitive Enhancement of Older People With Mild Cognitive Impairment (MCI) Living in the Community
Brief Title: Cognitive Training Using Feuerstein Instrumental Enrichment
Acronym: Feuerstein
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rambam Health Care Campus (Other)
Collaborators: Adolf und Mary Mil-Stiftung (Other); Helen Bader Foundation (Unknown); Montreal Jewish Community Fund (Unknown); Rochlin Family Foundation (Unknown)
Responsible Party: Principal Investigator, Tzvi Dwolatzky, Prof. Tzvi Dwolatzky, Rambam Health Care Campus
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: RMC_TD_23/2015
Record Dates: First submitted 2016-05-04; First posted 2016-05-17 (Estimated); Last update posted 2019-09-24 (Actual); Status verified 2019-09

CONDITIONS: Mild Cognitive Impairment
Keywords: older people; cognitive training
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Feuerstein Program (Active Comparator): The participants of the Intervention Group will participate in the Feuerstein mediated learning cognitive program.
  Interventions: Behavioral: Feuerstein Program
- Adler Program (Placebo Comparator): The Control Group will participate in the program of the Adler Institute dealing with social and emotional development without specific cognitive skills training.
  Interventions: Behavioral: Adler Program

INTERVENTIONS:
Behavioral: Feuerstein Program — Mediated learning cognitive enhancement program
  Arms: Feuerstein Program
Behavioral: Adler Program — Social and emotional group program
  Arms: Adler Program

SUMMARY:
Background: The Feuerstein Instrumental Enrichment Program was designed to prevent mental deterioration and preserve cognitive abilities among people aged 60 and above. The program is an applied practicable program based on the theories of Structural Cognitive Modifiability as well as on a Mediated Learning Experience. The program takes into consideration the unique characteristics and requirements of the older population. The program is composed of a variety of cognitive tasks that offer systematic activities intended to stimulate mental and cognitive development.

Objective: To examine the influence of the Feuerstein Program on the cognitive function and well-being of participants suffering from Mild Cognitive Impairment (MCI).

Hypothesis: The Feuerstein Program will improve cognitive abilities and functional well-being of the participants.

Methods: Residents of retirement homes will be offered to participate in the research. Participants will undergo cognitive and functional assessments that will be carried out on four specific dates. The participants of the Intervention Group will participate in the Feuerstein program using a method of mediated learning while the Control Group will participate in a program of the Adler Institute involving activities aimed at social and emotional development without specific cognitive skill training.

DETAILED DESCRIPTION:
Introduction

In recent decades, with the increase in life expectancy, the number of older people and their relative rate within the population have risen dramatically. This trend led to increased rates of people suffering from a mild cognitive disorder and dementia in developed countries. Mild Neurocognitive Disorder or Mild Cognitive Impairment (MCI) is defined as a transition state between successful aging and a state of dementia. This state is characterized by cognitive impairment and a decline in memory skills while daily functioning is maintained.

Older people diagnosed with MCI are at increased risk of developing dementia, particularly Alzheimer's disease. This risk is ranked at about 12% every year.

Since this is a pre-dementia stage, great importance lies in finding methods that could have prevented or at least decelerated the progress of MCI to dementia. Among the few effective programs are physical and cognitive activity.

The Feuerstein Program

This program is designated to prevent mental deterioration and preserve cognitive abilities among people aged 60 and above (hereinafter "The Feuerstein Program"). The program is the initiative and brainchild of Professor Reuven Feuerstein - Israel Prize Laureate, founder and President of the Feuerstein Institute for the Enhancement of Learning Potential.

The program is an applied practicable program based on the theories of Structural Cognitive Modifiability as well as on Mediated Learning Experience. For the needs of this program, the tools were suited to the unique characteristics and requirements of the elderly population.

The program is composed of a variety of tools (hereinafter: instrumental enrichment) that offer systematic activities intended to stimulate mental and cognitive development.

Instrumental enrichment is a set of tools dealing with required thinking skills and it is designated to significantly promote learning and thinking processes. The tasks of the various tools are free of educational content and they engage in pure learning and thinking processes. The tools are delivered through special mediation processes, for which teachers and supervisors are trained in specialized courses.

Objectives of the Feuerstein Program

The main objective: to enhance the transformation (variability) capacity of a human being.

The sub-objectives:

1. Correction and development of defective thinking skills, that are responsible for learning difficulties and the absence of transformation (variability).
2. Equipping the learner with literal and conceptual content that he requires during his learning processes.
3. Creating and establishing proper sound thinking and working habits.
4. Creating insight and awareness regarding the processes involved in learning.
5. Creating internal motivation for carrying out tasks.

The Learning Process

The instrumental enrichment tools are distributed to the participant as work sheets. The teacher creates a "mediating" dialogue between himself and the participants, thus enabling them to construct learning skills and essential thinking strategies. In addition, the teacher bridges the learning skills that were studied to the daily life of the elderly participant.

Products

1. Creating within them awareness to their learning and thinking processes (Metacognition) while introducing an optimistic and positive attitude towards the ability to effect a significant change in these areas.
2. Instill the elderly person with control over his thinking skills.
3. Enhancing the sense of capability of the elderly person.

The Intervention Focuses of the Instrumental Enrichment Tools that will be utilized in the Program

1. Methodical information gathering.
2. Orientation and function in space and time.
3. Comparison and sorting capabilities.
4. Memory.
5. Raising hypotheses and their examination.
6. Perspicuousness (clear wording) and naming capabilities.

The Control Group

The Control Group will participate in a program of the Adler Institute involving activities aimed at social and emotional development without specific cognitive skill training.

Research Objective

To examine the influence of the Feuerstein Program on the cognitive condition of participants suffering from Mild Cognitive Impairment (MCI).

Research Hypothesis

The Feuerstein Program will improve the cognitive and functional condition of the participants.

Methodology

Randomised controlled intervention study involving subjects with Mild Neurocognitive Disorder.

Research Assessment Tools

1. Cognitive screening by means of the MoCA (Montreal Cognitive Assessment) Test.
2. Instrumental daily function assessed by the Lawton and Brody's Instrument.
3. Depression screening based on the following question: "Are you feeling sad or depressed?". A positive response to this question has been found to be an efficient screening tool for depression.
4. Will to live based on the following question: If you could describe your will to live on a scale between 0 and 5, would you say that it is: 5 = very strong and 0 = no will to live.
5. CogSym (Cognitive Symptom) Meta-cognition questionnaire composed of ten items related to the cognitive ability of the examinee during his daily functioning. The examinee is asked to assess for each item, what is his ability level for the function being described, on a 5 levels scale (1 = excellent, 5 = inferior).
6. World Health Organization well-being index questionnaire.
7. The Neurotrax computerized cognitive assessment battery.

The intervention

Participants will be randomly allocated to an Intervention Group using the Feuerstein Program and a Control Group of the Adler Institute involving 30 twice weekly sessions each lasting 90 minutes over 15 weeks. Assessments will be performed at baseline, after session 15 and session 30, and finally at 6 months following study commencement.

Data Analysis The statistical analysis will be conducted as is customary in clinical research within the field.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 60 and above.
2. Hebrew/English speakers.
3. Expressing willingness to participate in the research and deliberately signing a consent form.
4. A diagnosis of MCI exists according to accepted clinical criteria - the examinee's score in the MoCA Test is within the range of 18-26 (inclusive).

Exclusion Criteria:

1. A medical or functional condition that will not allow the patient to participate in the intervention program within the research period.
2. Diagnosed patients suffering from depression, bipolar disorder or schizophrenia.
3. Patients who suffer from a diagnosed cognitive impairment other than MCI (delirium dementia or mental retardation).
4. Visual impairment that hasn't been amended by glasses.
5. Hearing impairment that hasn't been amended by a hearing aid.
6. Examinees whose MoCA Test's score is 17 and below or 27 and above.
7. Examinees who will receive the maximal score in one or more sections of the Lawton Test.
8. Examinees who will respond positively to a filter question regarding the topic of depression.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2015-09-03 (Actual); Primary Completion 2016-05-31 (Actual); Study Completion 2016-05-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline cognitive function | Through study completion, an average of 6 months
  Based on Neurotrax computerized neuropsychological assessment battery

CONTACTS AND LOCATIONS:
Overall Officials: Tzvi Dwolatzky, MD MBBCh, Principal Investigator — Rambam Health Care Campus
Locations (5):
- Israel (5):
  - Beit Yona, Beersheba
  - Ramat Tamir Retirement Home, Jerusalem
  - Beit Tovei Hair, Jerusalem
  - Bayit Balev Beit Ildan, Kiryat Motzkin
  - Bayit Balev Tel Aviv, Tel Aviv

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Carmel S. The will to live: gender differences among elderly persons. Soc Sci Med. 2001 Mar;52(6):949-58. doi: 10.1016/s0277-9536(00)00198-2. PMID 11234867
- [Background] Dwolatzky T, Whitehead V, Doniger GM, Simon ES, Schweiger A, Jaffe D, Chertkow H. Validity of a novel computerized cognitive battery for mild cognitive impairment. BMC Geriatr. 2003 Nov 2;3:4. doi: 10.1186/1471-2318-3-4. PMID 14594456
- [Background] Lifshitz M, Dwolatzky T, Press Y. Validation of the Hebrew version of the MoCA test as a screening instrument for the early detection of mild cognitive impairment in elderly individuals. J Geriatr Psychiatry Neurol. 2012 Sep;25(3):155-61. doi: 10.1177/0891988712457047. PMID 23124009
- [Background] Lachs MS, Feinstein AR, Cooney LM Jr, Drickamer MA, Marottoli RA, Pannill FC, Tinetti ME. A simple procedure for general screening for functional disability in elderly patients. Ann Intern Med. 1990 May 1;112(9):699-706. doi: 10.7326/0003-4819-112-9-699. PMID 2334082
- [Background] Topp CW, Ostergaard SD, Sondergaard S, Bech P. The WHO-5 Well-Being Index: a systematic review of the literature. Psychother Psychosom. 2015;84(3):167-76. doi: 10.1159/000376585. Epub 2015 Mar 28. PMID 25831962